CLINICAL TRIAL: NCT03006783
Title: Assessment of the Cross-face Nerve Graft in the Treatment of Facial Paralysis
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Tijn van Veen, M.M. van Veen, BSc, University Medical Center Groningen
Other Study IDs: TvanVeen
Record Dates: First submitted 2016-12-22; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Facial Palsy
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Cross-face nerve graft treated: People treated by a solitary cross-face nerve graft or in combination with another procedure.
  Interventions: Procedure: Cross-face nerve graft
- Hypoglossal-facial treated: People treated with a solitary hypoglossal-facial anastomosis.

INTERVENTIONS:
Procedure: Cross-face nerve graft — connecting the healthy facial nerve to the affected facial nerve
  Groups: Cross-face nerve graft treated

SUMMARY:
A retrospective and cross-sectional analysis of standard of care for facial paralysis involving the cross-face nerve graft in the past 20 years.

* Imagery analysis
* Questionnaires

DETAILED DESCRIPTION:
The investigators will retrospectively and cross sectionally analyze all patients treated with a cross-face nerve graft and another nerve transfer in our institution by image analysis and sending out quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Treated with one of the described procedures

Exclusion Criteria:

* Evaluation material present

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective cohort of people treated with a cross-face nerve graft or other nerve transfer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Symmetry of the mouth | March 2016 - October 2016
  Symmetry of the mouth expressed as the difference in millimeters between the position of the affected and the healthy corner of the mouth on a picture. An ideal symmetry would be 0 mm. Measured with the FACE-gram software.
Excursion of the mouth | March 2016 - October 2016
  Excursion of the mouth expressed as the difference in millimeters between the position of the affected corner of the mouth in repose and with smile on a picture. Measured with the FACE-gram software.
Disease-specific quality-of-life | March 2016 - October 2016
  A validated self-reported disease-specific quality-of-life questionnaire was used (Facial Clinimetric Evaluation scale). On which patients can score anything between 0 and 100 points (100 being healty).